CLINICAL TRIAL: NCT04756362
Title: Potential Impact in Clinical Practice of Early Exclusion Protocols for Acute Myocardial Infarction With High Sensitivity Troponin T in Different Scenarios (IN-HOspital Program to SystematizE Chest Pain Protocol-IN HOPE)
Brief Title: IN-HOspital Program to systematizE Chest Pain Protocol (IN-HOPE)
Acronym: In-Hope
Status: Completed | Type: Observational
Sponsor: Hospital Samaritano Paulista (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Pedro Gabriel Melo de Barros e Silva, Principal Investigator, Hospital Samaritano Paulista
Other Study IDs: 001/20
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chest Pain; Acute Coronary Syndrome
Keywords: Chest pain; Acute coronary syndrome; Troponin
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: A minimum of 294 patients will be included in the evaluation of 0 and 1 hour protocol (prospective evaluation).
- Retrospective cohort: A minimum of 1,000 patients will be included in the evaluation of prognostic value of high sensitive cardiac troponin < 5 ng/L(retrospective evaluation).

SUMMARY:
Multicenter Nationwide Study for Analysis of the Potential Impact in Clinical Practice of Early Exclusion Protocols for Acute Myocardial Infarction with High Sensitivity Troponin T

DETAILED DESCRIPTION:
Chest pain is the main clinical complaint in emergency room visits and represents the most common symptom of Acute Myocardial Infarction, which is the main cause of death in Brazil and worldwide. Although most patients with chest pain do not have a final diagnosis of AMI, they remain under observation until the diagnosis of AMI is excluded. The most current strategy recommended for rapid AMI exclusion uses high-sensitivity cardiac troponin T at time zero and one hour later. However, some points that have not yet been properly evaluated in previous studies can be evaluated in the current study:

* Evaluation of the early exclusion protocol (0 -1 hour) in a Brazilian population
* Evaluation of the early exclusion protocol (0 -1 hour) in isolation and associated with traditional risk scores (TIMI, GRACE, HEART and EDACS)
* Systematic evaluation of the early exclusion protocol (0 -1 hour) in patients without chest pain but with a pre-defined condition of suspected AMI
* Evaluation of the prognostic value of an isolated high-sensitivity cardiac troponin T < 5 ng/L in a diverse population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* The patient agrees and signs an informed consent form
* One of the following 2 criteria:

  1. Acute chest pain (last episode of pain beginning <6 hours after inclusion) or
  2. Syncope, dyspnea or epigastric pain without an obvious cause at the initial assessment (last episode of one of these symptoms beginning <6 hours after inclusion) associated with at least one of the following factors: Age ≥ 65 years, history of arterial disease, history of diabetes mellitus.

Exclusion Criteria:

* Cardiac arrest or hypoxemia or hemodynamic instability or cardioversion during the first hour of assessment
* Thrombolytic therapy, primary angioplasty or other medical condition that requires hospitalization identified within one hour after the evaluation
* Dialysis patients
* Patients with trauma
* Myocardial revascularization or acute myocardial infarction in the last month
* Pregnant and breastfeeding women
* Patient unable to be followed for 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with suspected acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 5497 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of early rule out for myocardial infarction diagnosis | 30 days
  Accuracy of the 0 and 1 hour algorithm using troponin for diagnosis of myocardial infarction compared to the gold standard with measurements every 3 hours

SECONDARY OUTCOMES:
Accuracy of early rule out for myocardial infarction according to type of symptoms | 30 days
  Accuracy of the 0 and 1 hour algorithm using troponin for diagnosis of myocardial infarction compared to the gold standard with measurements every 3 hours with or without chest pain
Accuracy of early rule out for myocardial infarction according to chest pain score (TIMI) | 30 days
  Accuracy of the 0 and 1 hour algorithm using troponin for diagnosis of myocardial infarction compared to the gold standard with measurements every 3 hours according to chest pain score (TIMI). TIMI score minimum 0 and maximum 7 points (higher scores mean a worse outcome).
Accuracy of early rule out for myocardial infarction according to chest pain score (EDACS) | 30 days
  Accuracy of the 0 and 1 hour algorithm using troponin for diagnosis of myocardial infarction compared to the gold standard with measurements every 3 hours according to chest pain score (EDACS). EDACS score minimum -6 and maximum +20 points (higher scores mean a worse outcome).
Accuracy of early rule out for myocardial infarction according to chest pain score (GRACE) | 30 days
  Accuracy of the 0 and 1 hour algorithm using troponin for diagnosis of myocardial infarction compared to the gold standard with measurements every 3 hours according to chest pain score (GRACE). GRACE score minimum 1 and maximum 372 points (higher scores mean a worse outcome).
Accuracy of early rule out for myocardial infarction according to chest pain score (HEART) | 30 days
  Accuracy of the 0 and 1 hour algorithm using troponin for diagnosis of myocardial infarction compared to the gold standard with measurements every 3 hours according to chest pain score (HEART). HEART score minimum 0 and maximum 10 points (higher scores mean a worse outcome).
Evaluation of the prognostic value (death and myocardial infarction within 30 days) of an isolated high-sensitivity cardiac troponin T < 5 ng/L in a diverse population. | 30 days
  Evaluation of the prognostic value (death and myocardial infarction within 30 days) of an isolated high-sensitivity cardiac troponin T < 5 ng/L in a diverse population (retrospective cohort).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Samaritano Paulista, São Paulo, Brazil

REFERENCES:
- [Derived] de Barros E Silva PGM, Ferreira AA, Malafaia F, Tavares Reis AFM, Sznejder H, Lopes Junior ACA, Agostinho CA, Fonseca LHO, Okitoi DVD, Correa CM, Zincone E, Cury MP, Rosa GAL, Ribeiro HB, Soeiro AM, de Oliveira CAL, Kuusberg GC, Ohe LN, Souza DO, Manfredi AB, Martins AF, Sampaio PPN, Vaz TB, Franco LF, Ferreira CEDS, Lopes RD; IN-HOPE Investigators. Potential performance of a 0 h/1 h algorithm and a single cut-off measure of high-sensitivity troponin T in a diverse population: main results of the IN-HOPE study. Eur Heart J Acute Cardiovasc Care. 2023 Nov 16;12(11):755-764. doi: 10.1093/ehjacc/zuad082. PMID 37450613